CLINICAL TRIAL: NCT05734677
Title: Emotion Regulation Group Intervention for Late Adolescents: a Clinical Trial
Brief Title: Emotion Regulation Group Study
Acronym: EmoReg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Camille Nemitz Piguet (Other)
Collaborators: Fondation Privée des HUG (Unknown)
Responsible Party: Sponsor-Investigator, Camille Nemitz Piguet, MD, PhD, PD, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-01883
Record Dates: First submitted 2023-01-11; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Emotional Dysfunction; Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- psychotherapeutic intervention with class risk A (low risk, no invasive procedure) (Experimental): an eight-week emotion regulation group intervention
  Interventions: Behavioral: Emotion regulation group

INTERVENTIONS:
Behavioral: Emotion regulation group — 90 minute sessions once a week for 8 weeks, in groups of eight participants. DBT, MBT and MBI inspired, psychoeducative intervention.

SUMMARY:
A clinical trial to evaluate the effects of an eight-week emotion regulation group intervention designed for adolescents (16-20 years old) on the levels of emotion dysregulation both self-reported by the adolescent and reported by his/her parent/caregiver (pre-post comparison). The long-term effect will also be measured at a third-time point, three months after the end of the intervention. The intervention will consist of 90-minute sessions once a week for 8 weeks, in groups of eight participants. The intervention proposed for this study is an adaptation from different interventions already in use for adolescents in clinical practice, such as Dialectical Behavior Therapy (DBT), Mentalization-Based Treatment (MBT) and Mindfulness-Based Intervention (MBI).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 16 to 20 years old.
* > 4 criteria of borderline symptoms (out of the 9 listed in the DSM-5) including emotional liability
* French speaking
* Availability during the whole study
* Willingness in participating to the intervention and the research
* Informed consent read and signed

Exclusion Criteria:

* Current hospitalization
* Psychotic disorder
* Severe and persistent substance addiction
* Antisocial personality disorder
* Inability to participate in group sessions
* Current pregnancy
* Non-French speaking
* Previous enrolment into the current study

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-09-06 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline in Difficulties in emotion regulation scale (DERS) | V2 (within two weeks after the end of the intervention)
  36 items self-report scale: Higher scores suggest greater problems with emotion regulation.
Changes from Baseline in Difficulties in emotion regulation scale (DERS) | V3 (3 months after the intervention)
  36 items self-report scale: Higher scores suggest greater problems with emotion regulation.
Changes from Baseline in Emotion Dysregulation Inventory (EDI) | V2 (within two weeks after the end of the intervention)
  Informant-report measure of emotion dysregulation
Changes from Baseline in Emotion Dysregulation Inventory (EDI) | V3 (3 months after the intervention)
  Informant-report measure of emotion dysregulation

SECONDARY OUTCOMES:
Changes from Baseline in Beck Depression Inventory (BDI-II) | V2 (within two weeks after the end of the intervention)
  Self-report inventory scored from 0 to 63 (higher score = more severe depressive symptoms)
Changes from Baseline in Beck Depression Inventory (BDI-II) | V3 (3 months after the intervention)
  Self-report inventory scored from 0 to 63 (higher score = more severe depressive symptoms)
Changes from Baseline in State-Trait Anxiety Inventory (STAI) | V2 (within two weeks after the end of the intervention)
  40 self-report items on a 4-point Likert scale: higher scores = greater anxiety
Changes from Baseline in State-Trait Anxiety Inventory (STAI) | V3 (3 months after the intervention)
  40 self-report items on a 4-point Likert scale: higher scores = greater anxiety
Changes from Baseline in self-report Family Attitude Scale (FAS) | V2 (within two weeks after the end of the intervention)
  30-item, Likert-scaled assessment for measuring the emotional climate of families (higher score = more critical family environment)
Changes from Baseline in self-report Family Attitude Scale (FAS) | V3 (3 months after the intervention)
  30-item, Likert-scaled assessment for measuring the emotional climate of families (higher score = more critical family environment)
Changes from Baseline in parent-report Family Attitude Scale (FAS) | V2 (within two weeks after the end of the intervention)
  30-item, Likert-scaled assessment for measuring the emotional climate of families (higher score = more critical family environment)
Changes from Baseline in parent-report Family Attitude Scale (FAS) | V3 (3 months after the intervention)
  30-item, Likert-scaled assessment for measuring the emotional climate of families (higher score = more critical family environment)
Changes from Baseline in Borderline Symptom List (BSL-23) | V2 (within two weeks after the end of the intervention)
  Self-rating tool for Borderline Personality Disorder (BPD) symptoms: higher scores = more likely to have BPD and associated challenges
Changes from Baseline in Borderline Symptom List (BSL-23) | V3 (3 months after the intervention)
  Self-rating tool for BPD symptoms: higher scores = more likely to have BPD and associated challenges
Changes from Baseline in self-report Strength & Difficulties Questionnaire (SDQ) | V2 (within two weeks after the end of the intervention)
  brief emotional and behavioural screening questionnaire assessing 25 attributes, some positive and others negative.
Changes from Baseline in self-report Strength & Difficulties Questionnaire (SDQ) | V3 (3 months after the intervention)
  brief emotional and behavioural screening questionnaire assessing 25 attributes, some positive and others negative.
Changes from Baseline in parent-report Strength & Difficulties Questionnaire (SDQ) | V2 (within two weeks after the end of the intervention)
  brief emotional and behavioural screening questionnaire assessing 25 attributes, some positive and others negative.
Changes from Baseline in parent-report Strength & Difficulties Questionnaire (SDQ) | V3 (3 months after the intervention)
  brief emotional and behavioural screening questionnaire assessing 25 attributes, some positive and others negative.
Changes from Baseline in Cognitive Emotion Regulation Questionnaire (CERQ) | V2 (within two weeks after the end of the intervention)
  Self-report measure designed to assess individual differences in cognitive regulation of emotions in response to stressful events. subscale scores can range from 4 to 20 with higher subscale scores indicating greater frequency of use of the specific cognitive strategy.
Changes from Baseline in Cognitive Emotion Regulation Questionnaire (CERQ) | V3 (3 months after the intervention)
  Self-report measure designed to assess individual differences in cognitive regulation of emotions in response to stressful events. subscale scores can range from 4 to 20 with higher subscale scores indicating greater frequency of use of the specific cognitive strategy.
Changes from Baseline in Kentucky inventory of mindfulness skills (KIMS) | V2 (within two weeks after the end of the intervention)
  self-report measuring Mindfulness on four scales: Observing, Describing, Act With Awareness, and Accept Without Judgment. Higher scores = higher mindfulness
Changes from Baseline in Kentucky inventory of mindfulness skills (KIMS) | V3 (3 months after the intervention)
  self-report measuring Mindfulness on four scales: Observing, Describing, Act With Awareness, and Accept Without Judgment. Higher scores = higher mindfulness
Changes from Baseline in Perceived Parental Autonomy Support Scale (P-PASS) | V2 (within two weeks after the end of the intervention)
  Measures parental autonomy-support and control of late adolescents and emerging adults. 24 items, assessed on a 7 point Likert scale.
Changes from Baseline in Perceived Parental Autonomy Support Scale (P-PASS) | V3 (3 months after the intervention)
  Measures parental autonomy-support and control of late adolescents and emerging adults. 24 items, assessed on a 7 point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Genève (HUG), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No